CLINICAL TRIAL: NCT01705964
Title: Intramuscular Epinephrine as an Adjunctive Treatment for Severe Pediatric Asthma Exacerbation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Kerry Caperell, Assistant Professor of Pediatrics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Caperell-Epi-001
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Asthma
Keywords: Status asthmaticus; Asthma exacerbation; Epinephrine; Adjunctive therapy
MeSH Terms: conditions — Asthma; Status Asthmaticus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IM epinephrine 1:1000 (Experimental): IM epinephrine 1:1000. The dose will be 0.2 mg for subjects 20-30 kg and 0.3 mg for subjects greater than 30 kg. This will be injected intramuscularly by an ED nurse into the anterior thigh muscles of the subject using a 1 ml syringe and a 23 gauge one inch needle.
  Interventions: Drug: IM epinephrine 1:1000
- No intervention (Sham Comparator): A sham band-aid will be applied to the anterior thigh of subjects who are randomized to the no intervention group.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: IM epinephrine 1:1000 — IM epinephrine 1:1000. The dose will be 0.2 mg for subjects 20-30 kg and 0.3 mg for subjects greater than 30 kg. This will be injected intramuscularly by an ED nurse into the anterior thigh muscles of the subject using a 1 ml syringe and a 23 gauge one inch needle.
  Arms: IM epinephrine 1:1000
Other: No intervention — A sham band-aid will be applied to the anterior thigh of subjects who are randomized to the no intervention group.
  Arms: No intervention

SUMMARY:
Project Aim: To determine if intramuscular epinephrine is an effective adjunct to inhaled bronchodilators (β2 agonists) for children with severe asthma exacerbation.

Hypothesis: IM epinephrine is an efficacious adjunct to inhaled bronchodilators (β2 agonists) for children with severe asthma exacerbation.

Intervention: Subjects will be randomly assigned (50% chance) to receive a weight based dose of IM epinephrine 1:1000 or no adjunctive medication. The dose will be 0.2 mg for subjects 20-30 kg and 0.3 mg for subjects greater than 30 kg. This will be injected intramuscularly by an ED nurse into the anterior thigh muscles of the subject using a 1 ml syringe and a 23 gauge one inch needle.

In addition to the study intervention, the standardized treatment pathway based on the current asthma guidelines in use at the investigator's center will be utilized. This pathway includes nebulized albuterol, ipratropium bromide, and systemic corticosteroids. The duration and dosages of these other interventions will be administered at the discretion of the treating provider.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 6 years and less than 18 years
2. Pre-existing diagnosis of asthma
3. Presenting to the ED with an asthma exacerbation

Exclusion Criteria:

1. History of chronic lung or upper airway disease other than asthma
2. History significant, uncorrected congenital heart disease or cardiac arrhythmia
3. History of thyroid disease
4. Impending respiratory failure
5. Allergy to epinephrine
6. Pregnancy
7. PEFR>60% of predicted and clinical asthma score less than 8

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2013-06; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Caperell, MD, Principal Investigator — University of Louisville
Locations (1):
- Kosair Children's Hospital, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IM Epinephrine 1:1000 | No Intervention
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM Epinephrine 1:1000 | No Intervention | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 24 | 49
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.00 (3.42) | 10.58 (2.76) | 10.29 (3.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 15 | 12 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 17 | 34
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Predicted Peak Expiratory Flow Rate (PEFR) at t15
Description: Change in percent of predicted Peak Expiratory Flow Rate (PEFR) 15 minutes after the study intervention (t15).
Time Frame: 15 minutes after the study intervention
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | IM Epinephrine 1:1000 | No Intervention
Number analyzed (Participants) | 25 | 24
percentage of predicted | 59.56 (17.11) | 52.45 (13.73)

2. Secondary Outcome: Disposition
Description: Disposition from the ED or rates of discharge.
Time Frame: At the time a dispostion from the ED is completed (usually within 4 hours of the study intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | IM Epinephrine 1:1000 | No Intervention
Number analyzed (Participants) | 25 | 24
Participants | 15 | 12

3. Secondary Outcome: Change in Percent of Predicted PEFR at t120
Description: Change in percent of predicted Peak Expiratory Flow Rate (PEFR) 120 minutes after study intervention compared to baseline
Time Frame: 120 minutes after the study intervention
Measure: Mean (Standard Deviation); unit: percentage of PEFR
Arm/Group | IM Epinephrine 1:1000 | No Intervention
Number analyzed (Participants) | 25 | 24
percentage of PEFR | 64.51 (21.68) | 56.18 (13.36)

4. Secondary Outcome: Breaths Per Minute at t120
Description: breaths per minute at t120 minutes compared to baseline
Time Frame: breaths per minute 120 minutes after the study intervention
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | IM Epinephrine 1:1000 | No Intervention
Number analyzed (Participants) | 25 | 24
breaths per minute | 24.29 (5.99) | 29.29 (7.96)

5. Secondary Outcome: Heart Rate at t120
Description: Heart rate at t120 minutes in beats per minute (BPM)
Time Frame: up to 120 minutes after the study intervention
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | IM Epinephrine 1:1000 | No Intervention
Number analyzed (Participants) | 25 | 24
Beats per minute | 147.65 (13.91) | 142.29 (16.30)

ADVERSE EVENTS:
Time Frame: 4 years 10 months
Arm/Group | IM Epinephrine 1:1000 | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-10-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT01705964/Prot_SAP_000.pdf